CLINICAL TRIAL: NCT06381596
Title: Retinal Fundus Flavoprotein Fluorescence in Age Related Macular Degeneration: New Insights From Multimodal Imaging
Brief Title: Retinal Fundus Flavoprotein Fluorescence in Age Related Macular Degeneration
Acronym: FPF in AMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2023-1715; A536000 (Other: UW- Madison); SMPH/OPHTHAL&VIS SCI/GEN (Other: UW- Madison); Protocol Version 11/26/2024 (Other: UW- Madison)
Record Dates: First submitted 2024-04-09; First posted 2024-04-24 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Geographic Atrophy; Age-Related Macular Degeneration
MeSH Terms: conditions — Geographic Atrophy; Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Fundus autofluorescence (FAF) imaging (Experimental)
  Interventions: Device: OcuMet Beacon

INTERVENTIONS:
Device: OcuMet Beacon — OcuMet Beacon is a novel fundus camera the can detect, capture, and assess FPF.

SUMMARY:
The goal of this clinical trial is to learn if the areas of stressed cells in the retina correlate to areas of disease identified in standard imaging and whether the images are helpful to identify potential areas of concern before symptoms or disease occurs. The main question it aims to answer is:

* to evaluate patterns of increased autofluorescence FPF in the setting of geographic atrophy

Participants will undergo FPF imaging using the OcuMet Beacon system.

DETAILED DESCRIPTION:
The goal of this clinical trial is to learn if areas of mitochondrial functional distress in the macula (as imaged using fundus flavoprotein fluorescence) correlate with areas of anatomic disease identified on standard fundus autofluorescence (FAF) imaging.

The study aims to evaluate patterns of anomalous fundus flavoprotein fluorescence (FPF) in patients with advanced geographic atrophy (GA) due to dry age-related macular degeneration.

Participants will undergo FPF imaging using the OcuMet Beacon system and FAF imaging using Heidelberg Spectralis.

ELIGIBILITY:
Inclusion Criteria:

* 50 years or older and may be either male or female of any race
* Established diagnosis of GA due to AMD
* GA characteristics: GA area of between 1.25 mm² and 23 mm², with seventy percent of eyes having GA area ranging from 2.5 mm2 to 17.5 mm2. GA may be unifocal or multifocal. GA may be subfoveal or extrafoveal, with twenty-five percent of eyes having subfoveal GA. The presence of concurrent peripapillary atrophy will not exclude subjects from participation
* Willing to participate as evidenced by signing the written informed consent

Exclusion Criteria:

* Unable to tolerate ophthalmic imaging
* Presence of neovascular AMD on OCT as confirmed by an ophthalmologist
* Presence of significant media opacity preventing adequate retinal imaging
* Presence of concurrent retinal disease which may confound assessment

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2024-04-16 (Actual); Primary Completion 2025-05-27 (Actual); Study Completion 2025-05-27 (Actual)

PRIMARY OUTCOMES:
Limits of agreement between the fundus autofluorescence (FAF) area of GA images taken with the Heidelberg Spectralis to the flavoprotein fluorescence (FPF) area of GA with images taken with the OcuMet Beacon | Up to 45 minutes
  The equivalence test will be performed using the estimated fixed effect coefficient and standard errors derived from the mixed-effects model, where the null hypothesis is that the difference in measurements between the two devices is outside the equivalence bounds of -2.5% to 2.5%.

SECONDARY OUTCOMES:
Compare the cross-sectional associations between FPF intensity (average pixel intensity over a 5.5 mm-diameter region centered at the macula) to FAF area at the time of measurement | Up to 45 minutes
Compare the cross-sectional associations between best corrected visual acuity (BCVA - using Early Treatment Diabetic Retinopathy Study, greater number of letters read correctly equals better vision) to FAF area at the time of measurement | Up to 45 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Mihai Mititelu, MD, MPH, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- Department of Ophthalmology and Visual Sciences, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No